CLINICAL TRIAL: NCT06291610
Title: Feasibility Testing a Decision-support Intervention for Clinical Trials
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Aarhus University Hospital
Record Dates: First submitted 2024-02-08; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Head and Neck Neoplasms
Keywords: Clinical trial decision making; Patient involvement; Decision coaching; Feasibility study; Complex intervention
MeSH Terms: conditions — Head and Neck Neoplasms; Patient Participation

STUDY DESIGN:
Intervention Model Description: Pre- and post-intervention measures in two consecutive groups.
Masking Description: Patients are recruited anonymous
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decision intervention group (Other): The decision intervention will be tested in one arm (group)
  Interventions: Behavioral: Clinical trial decision support intervention

INTERVENTIONS:
Behavioral: Clinical trial decision support intervention — 1. a patient decision aid tailored to clinical trial participation
  2. decision coaching consultations carried out by trained healthcare professionals.
  3. a training program in decision coaching will be an integrated part of the intervention.

SUMMARY:
A decision-support intervention are developed for a Danish nationwide randomised controlled trial (RCT) among patients with laryngeal and pharyngeal cancer referred to curative intended radiotherapy. The primary endpoints in this RCT are levels of dysphagia and xerostomia.

The decision-support intervention consists of three components, including (1) a patient decision aid tailored to clinical trial participation and (2) decision coaching consultations carried out by trained healthcare professionals. Finally, (3) a training program in decision coaching will be an integrated part of the intervention.

To feasibility test (beta test) the intervention, 60 patient participants will be included, separated into pre- (n=30) and post- (n=30) intervention groups. Pre-intervention to complete the survey based on current clinical practice. Post-intervention to complete the survey following engagement in the decision support intervention.

A total of 12 physicians will be recruited and trained in decision coaching. To assess the acceptability of the intervention, the physicians will be interviewed. Additionally, they will be asked to audio-record two decision coaching sessions to test the fidelity of the intervention.

DETAILED DESCRIPTION:
Decision-support interventions for patients considering clinical trial participation may promote informed decisions. However, decision interventions for people considering clinical trial participation are still limited.

This study aims to develop and test the acceptability and feasibility of a decision-support intervention to enhance informed decision-making regarding clinical trial participation.

A decision-support intervention has been developed for a Danish nationwide randomised controlled trial (RCT) among patients with laryngeal and pharyngeal cancer referred to curative intended radiotherapy. The primary endpoints in this RCT are levels of dysphagia and xerostomia.

The decision-support intervention consists of three components, including (1) a patient decision aid tailored to clinical trial participation and (2) decision coaching consultations carried out by trained healthcare professionals. Finally, (3) a training program in decision coaching will be an integrated part of the intervention.

To feasibility test (beta test) the intervention, 60 patient participants will be included, separated into pre- (n=30) and post- (n=30) intervention groups. Pre-intervention to complete the survey based on current clinical practice. Post-intervention to complete the survey following engagement in the decision support intervention.

A total of 12 physicians will be recruited and trained in decision coaching. To assess the acceptability of the intervention, the physicians will be interviewed. Additionally, they will be asked to audio-record two decision coaching sessions to test the fidelity of the intervention.

Methods:

Patient participants outcome ( questionnaire survey)

1. The stages of decision making measure (self translated forward/backward)
2. Decisional conflict scale
3. The decision preparation scale (post intervention measure)
4. Items on health literacy related to the specific context (understanding the trial, the treatment modalities, practical issues, etc.)
5. Decision preference

The interviews with the clinicians (decision coaches) will follow the interpretive description methodology and be conducted as qualitative, semi-structured audio-recorded interviews. The interviews will be carried out on the telephone.

The quantitative data will be hosted, organised, and analysed in STATA. The qualitative data will be hosted, organised, and analysed in a software system called NVivo.

To evaluate the impact of the decision-support intervention, it is necessary to assess the extent to which it is used as intended in clinical practice. This is referred to as a fidelity test. Hence, the decision coaches will be provided with dictaphones and asked to audio-record the consultations. The audio records will be evaluated using the Decision Support Analysis Tool (DSAT-10), which is a tool to assess practitioners' use of decision support and communication skills during a clinical encounter.

Further studies

Building upon the current study, the potential for further development, implementation and evaluation across proton therapy clinical trials will be determined.

Assessing a decision support intervention for trial participation in a single host trial is challenging due to the limited period of the host trial and insufficient statistical power for comparative tests.

Additional intervention development could involve establishing an online decision support intervention platform for Danish proton therapy clinical trials and a training platform in decision coaching for healthcare professionals. Moreover, integrating measurements (decisional conflict, etc.) as active pro measures to identify decisional needs during decisional coaching could be explored.

A cluster randomised trial is the most suitable approach for full-scale implementation and evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer of the pharynx or larynx
* Received verbal information regarding DAHANCA 35
* Read the patient information folder from DAHANCA 35
* Above 18 years
* Danish speaking

Exclusion Criteria:

* Dyslexia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Decisional conflict scale | The day of signing the clinical trial consent form
  Measures the level of patients decisional conflict
The decision preparation scale | The day of signing the clinical trial consent form
  Measures patients ability to prepare for decision-making

SECONDARY OUTCOMES:
The stages of decision making measure | The day of signing the clinical trial consent form
  Measures the stage patients are in during the decision-making process
Items on health literacy | The day of signing the clinical trial consent form
  Related to the specific context (understanding the trial, the treatment modalities, practical issues, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Anne W Kristensen, MSc, Study Chair — Aarhus University Hospital; Cai W Grau, Professor, Study Director — Aarhus University Hospital; Jeppe Friborg, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No